CLINICAL TRIAL: NCT05761054
Title: Sarcoma Preoperative Radiation With Simultaneous INTegrated Boost (SPRINT)
Acronym: SPRINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Professor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPRINT
Record Dates: First submitted 2023-02-13; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Soft Tissue Sarcoma
Keywords: soft tissue sarcoma (STS); Intensity Modulated Radiotherapy (IMRT); boost; radiotherapy; locally advanced soft tissue sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A (Experimental)
  Interventions: Radiation: RT

INTERVENTIONS:
Radiation: RT — The treatment will be administered in 25 daily fractions (Monday-Friday) at the disease site to include the region of suspected micrometastatic spread (Clinical Target Volume 1, CTV1) at a dose of 50 Gy (2Gy
  / fraction) with SIB intensification on volume reduced corresponding to the interface sites between the tumor and the vascular / nerve axes (Clinical Target Volume 2, CTV2) at a dose of 60 Gy (2.4 Gy / fraction). The association with neoadjuvant chemotherapy based on anthracyclines is allowed.

SUMMARY:
Intervention prospective monocentric one arm study on the use of neoadjuvant radiotherapy with simultaneous integrated boost (Simultaneous Integrated Boost, SIB) in patients with STS with indication for preoperative radiotherapy. The treatment will be administered in 25 daily fractions (Monday-Friday) at the disease site to include the region of suspected micrometastatic spread (Clinical Target Volume 1, CTV1) at a dose of 50 Gy (2Gy

/ fraction) with SIB intensification on volume reduced corresponding to the interface sites between the tumor and the vascular / nerve axes (Clinical Target Volume 2, CTV2) at a dose of 60 Gy (2.4 Gy / fraction). The association with neoadjuvant chemotherapy based on anthracyclines is allowed.

DETAILED DESCRIPTION:
Intervention prospective monocentric one arm study on the use of neoadjuvant radiotherapy with simultaneous integrated boost (Simultaneous Integrated Boost, SIB) in patients with STS with indication for preoperative radiotherapy. The treatment will be administered in 25 daily fractions (Monday-Friday) at the disease site to include the region of suspected micrometastatic spread (Clinical Target Volume 1, CTV1) at a dose of 50 Gy (2Gy

/ fraction) with SIB intensification on volume reduced corresponding to the interface sites between the tumor and the vascular / nerve axes (Clinical Target Volume 2, CTV2) at a dose of 60 Gy (2.4 Gy / fraction). The association with neoadjuvant chemotherapy based on anthracyclines is allowed. Objective: The primary objective is to evaluate the benefit of radiotherapy with partial simultaneous integrated boost to the area at risk of incomplete resection in the neoadjuvant treatment of soft tissue sarcoma candidate for conservative surgery. The secondary objectives are to evaluate the outcomes and toxicity Study population: Patients with de novo or locoregional recurrence of STS after surgery.

Estimated enrollment: 33 Inclusion criteria: STS candidate for surgical resection; age > 18 years Exclusion criteria: previous radiotherapy over the region of interests, inability to express informed consent; planned amputation. Study arm: Intensity Modulated Radiotherapy Study duration: 2 years Enrollment period: 3 years Global study duration: 5 years Current primary outcomes measures: Oncologically negative resection rate (R0 rate) Current secondary outcomes measures: Pathologic Complete Response rate (pCR); Overall Survival (OS); Disease Specific Survival (DSS) Local-Relapse Free Survival (LRFS); Distant-Metastases-Free Survival (DMFS); incidence of acute and late toxicity according to CTCAE v5.0 classification

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Confirmed histological diagnosis of soft tissue sarcoma
* Candidate for conservative surgery
* Performance status ≤ 1 according to WHO (or ≥ 70 according to KPS) before starting the treatment in the office.

Exclusion Criteria:

* Previous radiotherapy at the same site
* Candidate for Surgical Amputation
* Patients with comorbidities for collagen diseases
* Psychiatric disorders that may preclude obtaining the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
R0 rate | immediately after surgery
  Oncologically negative resection rate

SECONDARY OUTCOMES:
(pCR); | immediately after surgery
  Pathologic Complete Response rate
(OS); | through study completion, average of 36 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: lorenzo livi, Dr, Principal Investigator — AOU Careggi
Locations (1):
- AOU Careggi, Florence, Fi, Italy

IPD SHARING:
Plan to Share IPD: Yes